CLINICAL TRIAL: NCT01810133
Title: Retrospective Data Analysis: Evaluation of Co-morbidity Scales in Peri-operative Medicine
Brief Title: Evaluation of Co-morbidity Scales
Acronym: Ko-MoSkau
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charite University, Berlin, Germany
Other Study IDs: Ko-MoSkaU
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Mortality
Keywords: Comorbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anesthesia patients: All patients undergoing general anesthesia between January 2006 and December 2011 in Charité - University Berlin

SUMMARY:
Peri-operative mortality depends on the patient's co-morbidities. ASA Physical Status (American Society of Anesthesiology) is the most commonly scale to assess this parameter and has yet been repeatedly criticized in the past for its discriminatory power.

Few studies have shown both the ASA physical status and the more detailed and more time-consuming Charlson Comorbidity Index to be equivalent in certain patient populations.

The purpose of this observational study is to compare the predictive value of both scales with regards to all-cause in-hospital mortality and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1) All male and female Patients who underwent anesthesia within the study time period (January 2006 and December 2011) in the Charité - University Berlin, Department of Anesthesiology and Intensive Care Medicine CVK/CCM.

Exclusion Criteria:

None

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing general anesthesia between January 2006 and December 2011
Sampling Method: Probability Sample
Enrollment: 230034 (Actual)
Dates: Start 2006-01; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of patients that died after surgery during their hospital stay | 1 year
  Electronic patient charts are revised for the complete hospital length of stay for co-morbidities, intra-operative data and post-operative all-cause in-hospital mortality.

SECONDARY OUTCOMES:
Hospital length of stay associated with surgery | 1 year
  Electronic patient charts are revised for the complete hospital length of stay for co-morbidities, intra-operative data and post-operative all-cause in-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, CVK and CCM, Charité-University, Berlin, Germany, Germany